CLINICAL TRIAL: NCT06076720
Title: Evaluation of New Head-mounted Visual Aids Among Patients With Low Vision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ123
Record Dates: First submitted 2023-09-24; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Glaucoma; Age-related Macular Degeneration; Retinitis Pigmentosa; Diabetic Retinopathy
Keywords: Visual rehabilitation of low vision, head-mounted devices
MeSH Terms: conditions — Glaucoma; Macular Degeneration; Retinitis Pigmentosa; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New head-mounted visual aids (Experimental): Wearing different head-mounted visual aids
  Interventions: Device: New head-mounted visual aids

INTERVENTIONS:
Device: New head-mounted visual aids — New head-mounted visual aids such as Beyes, HOLA, Acesight and OXSIGHT are the latest wearable electronic visual aids

SUMMARY:
Glaucoma, age-related macular degeneration (AMD), retinitis pigmentosa, RP, diabetic retinopathy (DR) are the most common blinding eye diseases in the world. Vision and visual field are often severely impaired, quality of life is reduced, and personal and family burdens are heavy. This kind of low vision people, can use visual AIDS and other instruments for visual rehabilitation training, maximize the function of residual vision, improve the quality of life. Beyes, HOLA, Acesight and OXSIGHT are among the latest eyeglasses devices that are expected to improve the quality of life for people with low vision. This research group intends to recruit advanced patients with primary glaucoma, AMD, RP, DR and other common blinding eye diseases who visited Zhongshan Ophthalmology Center of Sun Yat-sen University from June 2021 to December 2022 to study the changes of visual function and quality of life after wearing this new type of head-worn visual aids, and analyze relevant factors combined with clinical data. To evaluate the effect and influencing factors of the new head-mounted visual AIDS on patients, and provide theoretical basis for subsequent clinical research.

DETAILED DESCRIPTION:
1. Low vision Low visual acuity refers to a patient who has functional impairment of vision even after treatment or standard refractive correction. The visual acuity of the good middle eye in both eyes is less than 0.3, or the field radius is ≤20°, but still has the ability to use the remaining vision to perform a certain visual activity. In China, low vision caused by eye diseases (such as glaucoma, AMD, RP, DR) can lead to behavioral loss of patients, and standardized rehabilitation treatment of low vision can help 90% of visual impairment patients improve the utilization rate of residual vision, becoming an important way to compensate for the loss of visual function of this group.
2. Visual rehabilitation of low vision The latest definition of visual rehabilitation is a kind of multidisciplinary comprehensive rehabilitation therapy. By ophthalmologists, depending on the light, low vision devices, low vision rehabilitation counselors professional therapists, social workers and psychologists of the multidisciplinary team, using physical, audio, electronic, optical instruments, and life skills training, help patients with low vision to use its residual vision and development skills available to offset the impact of visual impairment in patients, To improve their self-living ability and quality of life. There are three treatment levels: discovery, guidance and referral; Individual rehabilitation; Multidisciplinary visual rehabilitation.

   The first step of visual rehabilitation is often accurate optometry in order to obtain the best corrected vision, which is also an important basis for the success of visual rehabilitation. On the basis of refractive correction, it can obviously improve the daily living ability and quality of life of the patients with low vision by providing them with appropriate visual aids and corresponding training of using visual aids. Visual aids are generally divided into near-use and far-use visual aids, in which near-vision and reading ability are the focus of functional vision assessment and rehabilitation. Traditional used visual aids have hand-held magnifier, vertical magnifier, glasses and electronic visual aids. Compared with optical visual aids, electronic visual aids have the advantages of clear imaging, adjustable magnification and contrast.
3. Research status of smart wearable devices Traditional visual AIDS achieve the effect of object image amplification through the principle of optics, but have fixed magnification rate, reduced field of vision, small depth of field, short working distance, can not adjust the contrast and other shortcomings. In recent years, video wearable devices have been gradually applied in the field of visual rehabilitation, with the advantages of adjustable magnification, adjustable contrast and high clarity, overcoming the limitations of traditional optical devices, including eSight 3, NuEyes, IrisVision, etc.

Currently, there are few studies on wearable electronic visual aids. Walter Wittich et al. conducted an intervention trial on 51 patients with low vision and confirmed that wearable electronic visual aids can improve patients' visual acuity, spatial object recognition ability, and reading and activity ability. In the study of middle-advanced glaucoma, Yogesh Patodia et al. found that wearable electronic visual aids can also improve their long-range and near-range vision.

Smart glasses such as Beyes, HOLA, Acesight and OXSIGHT are the latest wearable electronic visual aids to hit the market, featuring advantages of lighter weight, comfortable wearing, better imaging quality and multi-mode assisted visual recognition. However, the effect and influencing factors of this kind of smart glasses on advanced patients with glaucoma, AMD, RP, DR and other common blinding eye diseases are still unclear, which requires further exploration by researchers.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥10 years, able to complete all tests and inspections
2. a definite diagnosis of low vision or blindness:

   * Criteria for low vision: the best corrected visual acuity of the better eye ≤0.3, and ≥0.05 or the visual field of the better eye no greater than 20° in radius around central fixation

     * Criteria for blindness: the best corrected visual acuity of the better eye <0.05 or the visual field of the better eye no greater than 10° in radius around central fixation
3. Visual acuity, intraocular pressure, and other eye conditions have been stable for more than 6 months.

Exclusion Criteria:

1. unable to cooperate with related inspections
2. a history of eye surgery or eye laser within six months
3. serious systemic diseases, such as neurological diseases, cardiovascular diseases, psychological diseases, malignant tumors, etc.
4. pregnant or lactating women
5. those who refuse to sign the informed consent or voluntarily withdraw from the study due to discomfort or other reasons.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes in the Glaucoma Visual Functioning Questionnaire-40 (GVFQ-40) scores at different time points | 8 weeks after intervention
  The GVFQ-40 consists of 40 items and measures the difficulty of daily activities of glaucoma patients in five domains of functioning (mobility, visual tracking, reading, identification and night vision ). Each item has six answer options, that is, no difficulty (score = 1), mild difficulty (score = 2), moderate difficulty (score = 3), extremely difficult (score = 4), completely unable to complete (score = 5), and do not perform for nonvisual reasons (no score). The GVFQ-40 was administered at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.
Comparison of changes in the National Eye Institute-Visual Function Questionnaire-25 (NEI VFQ-25) scores at different time points | 8 weeks after intervention
  The National Eye Institute-Visual Function Questionnaire-25 (NEI VFQ-25) is a valid and reliable vision-related quality of life (QOL) questionnaire designed for persons who have chronic eye diseases or low vision. It includes 25 items that comprise 11 subscales on different aspects of vision-related functioning and QOL and 1 item on general health. NEI VFQ-25 scores range from 0 to 100, with a higher score representing better functioning. The NEI VFQ-25 was administered at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.
Comparison of changes in the Low Vision Quality-of-Life Questionnaire (LVQOL) scores at different time points | 8 weeks after intervention
  The Low Vision Quality-of-Life Questionnaire (LVQOL) specifically examines the QOL of patients with visual disability. The LVQOL is of the latter type, with the 25 items producing a summed score between 0 and 125 (the higher the score, the higher the quality of life). The 25 items are grouped into 4 subscales: distance vision, mobility and lighting; adjustment; reading and fine work; and daily life activities. As a convenient tool, LVQOL is widely used in clinical settings to evaluate effects of clinical treatment and corresponding strategies of low-vision rehabilitation. The LVQOL was tested at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.

SECONDARY OUTCOMES:
Comparison of changes in visual acuity at different time points | 8 weeks after intervention
  Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart was used. The examination was performed at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.
Comparison of changes in contrast sensitivity at different time points | 8 weeks after intervention
  Pelli-Robson Contrast Sensitivity Charts were used. The examination was performed at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.
Comparison of changes in kinetic visual field at different time points | 8 weeks after intervention
  Kinetic visual field was measured by the automated perimetry. The examination was performed at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.
Comparison of changes in functional magnetic resonance imaging (MRI) at different time points | 6 months after intervention
  The whole brain BOLD and T1 structures were scanned using a MAGNETOM Verio 3 T MR scanner. Structural and functional MRI scans were performed at baseline and at 1 week, 8 weeks, and 6 months after intervention.
Comparison of changes in mobility test at different time points | 8 weeks after intervention
  A mobility test was performed to evaluate patients' functionality in 2 scenarios: using their presenting distance visual acuity with no aids and using the head-mounted aids. A loop-shaped obstacle course consisting of stationary obstacles from floor to head level was designed for this test. The test was performed at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.
Comparison of changes in visual scanning test at different time points | 8 weeks after intervention
  A visual scanning test was performed to evaluate patients' functionality in 2 scenarios: using their presenting distance visual acuity with no aids and using the head-mounted aids. Four pictures were designed for this test. Each picture involved seven types of randomly aligned figures and the four patterns of pictures with different alignments were prepared to determine the scores of individuals and the time required to answer. The test was performed at baseline and 1 day, 1 week, 4 weeks, and 8 weeks after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fontenot JL, Bona MD, Kaleem MA, McLaughlin WM Jr, Morse AR, Schwartz TL, Shepherd JD, Jackson ML; American Academy of Ophthalmology Preferred Practice Pattern Vision Rehabilitation Committee. Vision Rehabilitation Preferred Practice Pattern(R). Ophthalmology. 2018 Jan;125(1):P228-P278. doi: 10.1016/j.ophtha.2017.09.030. Epub 2017 Nov 4. No abstract available. PMID 29108747
- See also: Vision Rehabilitation Preferred Practice Pattern® — https://pubmed.ncbi.nlm.nih.gov/29108747/